CLINICAL TRIAL: NCT02644863
Title: Phase II Clinical Study of Patients Randomized, Open, Controlled Evaluation of Autologous Tumor Tissue Antigen Sensitized DC-CIK Cells Combined With Chemotherapy in the Treatment of Patients With Esophageal Resection
Brief Title: Autologous Tumor Tissue Antigen-sensitized DC-CIK Cells Combined With Chemotherapy for Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Hornetcorn Bio-technology Company, LTD (Industry)
Collaborators: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYK-esophageal cancer
Record Dates: First submitted 2015-12-28; First posted 2016-01-01 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2015-12

CONDITIONS: Esophageal Neoplasms; Neoplasms; Digestive System Neoplasms; Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Neoplasms; Digestive System Neoplasms | interventions — Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DC-CIK (Experimental): After accepting chemotherapy according to guidelines,patients will receive 3 cycles of autologous DC-CIK treatment.
  Interventions: Drug: Paclitaxel; Biological: DC-CIK; Drug: Cisplatin
- Chemotherapy (Sham Comparator): After the Chemotherapy by Paclitaxel and Cisplatin, patients will just regularly follow up.
  Interventions: Drug: Paclitaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel 175mg/m2 IV over 2 hours,day 1; Repeat every 3 weeks;regimen for 3 cycles
  Other Names: TP
Biological: DC-CIK — Antigen-sensitized DC-CIK 8×10^9 autologous tumor lysate pulsed D-CIK cells for each infusion, IV (in the vein) for 3 cycles, each cycle received four infusions on day 14, 16, 30 and 32.
  Arms: DC-CIK
Drug: Cisplatin — Cisplatin 30mg/m2 IV on 1-3 days, Repeat every 3 weeks;regimen for 3 cycles

SUMMARY:
This study evaluates the safety and efficacy of D-CIK immune cells combined with chemotherapy after resection of esophageal cancer

DETAILED DESCRIPTION:
60 patients of esophageal cancer with TNM stage of tumor stage II-III,who had received surgery and kept their tumor tissue, will be randomly divided into group A (receive cancer tissue antigen sensitized D-CIK immune cells in combination with chemotherapy treatment) or group B (just receive chemotherapy), and the randomize ratio will be 1:1. Patients in group A will receive 3 cycles of autologous antigen-sensitized DC-CIK cells treatment (every 4 weeks) and chemotherapy. Patients in group B will receive only 3 cycles chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old;
* Clinical diagnosis of esophageal cancer patients,tumor TNM stageII-III;
* Patients who can accept curative operations;
* Patients who have a life expectancy of at least 3 months; .Eastern Cooperative Oncology Group (ECOG) performance status was 0-2.

Exclusion Criteria:

* White blood cell <3 x 10^9/L,Platelet count <75 x 10^9/L;BUN and Cr more than normal limits on 3.0 times ;
* Known or suspected allergy to the investigational agent or any agent given in association with this trial;
* Pregnant or lactating patients;
* Known history of Human Immunodeficiency Virus (HIV), Hepatitis C Virus (HCV) or TreponemaPallidun (TP) infection;
* Patients who are suffering from serious autoimmune disease;
* Patients who had used long time or are using immunosuppressant;
* Patients who had active infection;
* Prior use of any anti-cancer treatment in 30 days;
* Now or recently will join another experimental clinical study ;
* History of organ allograft;
* Other situations that the researchers considered unsuitable for this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 years
  The time of randomization begins to cause the death of any cause

SECONDARY OUTCOMES:
Progress-free survival | 3 years
  The time of randomization begins to tumor progression
Quality of life (QOL) | 3 years
  Assess the quality of life of patients
Phenotypic analysis of T cells | 1 year
  The number of CD3+ (or CD8+ or CD4+ or CD56+) T cell

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyuan Wang, Professor, Study Chair — Affiliated Tumor Hospital of Guangzhou Medical University Immunotherapy center
Locations (1):
- Affiliated Tumor Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided